CLINICAL TRIAL: NCT00001748
Title: HLA-Mismatched Peripheral Blood Mobilized Hematopoietic Precursor Cell Transplantation for Hematological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980122; 98-H-0122
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-08

CONDITIONS: Graft vs Host Disease; Hematologic Neoplasms; Lymphoma; Myelodysplastic Syndromes; Myeloid Leukemia
Keywords: Cyclophosphamide; Donor Apheresis; Graft vs. Host Disease; Graft-Versus-Leukemia; Leukemic Relapse; Myeloma; Peripheral Blood Stem Cells; Whole Body Irradiation; Acute Lymphoblastic Leukemia (ALL); Chronic Lymphocytic Leukemia (CLL); Chronic Myelogenous Leukemia (CML); Hematological Malignancies; Myelodysplastic Syndrome; Myeloproliferative Disorders
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms; Lymphoma; Myelodysplastic Syndromes; Leukemia, Myeloid; Neoplasms, Plasma Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myeloproliferative Disorders

INTERVENTIONS:
Procedure: Peripheral blood progenitor cell transplant

SUMMARY:
Many patients with hematological malignancies potentially curable by bone marrow transplantation are not considered for transplantation because an HLA identical family or unrelated donor is unavailable. For these patients the only curative option is a transplant from a partially matched family donor. Such transplants are feasible but are less successful than matched sibling donor transplants. The main problems with mismatched transplants are graft rejection, graft-vs-host disease, and regimen-related mortality. This restricts the use of mismatched transplants to patients less than 45 years at high risk of dying from the hematological malignancy.

This protocol evaluates a new preparative regimen designed to ensure stem cell engraftment by increased immunosuppression, followed by a G-CSF mobilized T cell depleted, stem cell rich, peripheral blood progenitor cell (PBPC) transplant from a mismatched related donor in patients with high risk hematological malignancies.

This phase I study evaluates engraftment and GVHD following T cell depleted, HLA-mismatched PBPC transplants. Stopping rules will be used to make modifications to the protocol in the event of graft failure.

The end points of the study are graft take, acute and chronic GVHD, leukemic relapse, transplant-related mortality, death and leukemia-free survival. Patients will be followed up for 5 years. It is planned to treat up to 35 patients aged between 10 and 45 years.

DETAILED DESCRIPTION:
Many patients with hematological malignancies potentially curable by bone marrow transplantation are not considered for transplantation because an HLA identical family or unrelated donor is unavailable. For these patients the only curative option is a transplant from a partially matched family donor. Such transplants are feasible but are less successful than matched sibling donor transplants. The main problems with mismatched transplants are graft rejection, graft-vs-host disease, and regimen-related mortality. This restricts the use of mismatched transplants to patients less than 45 years at high risk of dying from the hematological malignancy.

This protocol evaluates a new preparative regimen designed to ensure stem cell engraftment by increased immunosuppression, followed by a G-CSF mobilized T cell depleted, stem cell rich, peripheral blood progenitor cell (PBPC) transplant from a mismatched related donor in patients with high risk hematological malignancies.

This phase I study evaluates engraftment and GVHD following T cell depleted, HLA-mismatched PBPC transplants. Stopping rules will be used to make modifications to the protocol in the event of graft failure.

The end points of the study are graft take, acute and chronic GVHD, leukemic relapse, transplant-related mortality, death and leukemia-free survival. Patients will be followed up for 5 years. It is planned to treat up to 35 patients aged between 10 and 45 years.

ELIGIBILITY:
Patient:

Ages 10-45 years.

Chronic myelogenous leukemia, any of these categories: accelerated phase or blast transformation.

Acute lymphoblastic leukemia, any of these categories: Adults (greater than 18 years) in any remission with high-risk features (presenting leukocyte count greater than 100,000/cu mm, Karyotypes t9; 22, t4, t19, t11, biphenotypic leukemia). All second remissions, primary induction failure including partial remission, partially responding or untreated relapse.

Acute myelogenous leukemia (AML): All AML in second or subsequent remission, primary induction failure or partial remission and resistant relapse.

Myelodysplastic syndromes, any of these categories: refractory anemia with excess of blasts, transformation to acute leukemia, chronic myelomonocytic leukemia.

Myeloproliferative disorders undergoing transformation to terminal stages.

Chronic lymphocytic leukemia (CLL) in Richter transformation.

High-grade lymphoma, refractory to standard treatment approaches, mantle cell lymphoma.

No major organ dysfunction precluding transplantation.

DLCO greater than 65% predicted.

Left ventricular ejection fraction: greater than 40% predicted.

ECOG performance status of 0 or 1.

Informed consent given. Informed consent from parents for minors.

Women of childbearing age with a negative pregnancy test may participate.

Donor:

Partially HLA matched family donor (3-5/6 matches).

Fit to receive G-CSF and give peripheral blood stem cells (normal blood count, normotensive, and no history of stroke).

Informed consent given.

Patients or donors must not be pregnant or nursing.

Must not have ECOG performance status of 2 or more.

No severe psychiatric illness in patient or donor: Mental deficiency sufficiently severe as to make compliance with the BMT treatment unlikely and making informed consent impossible.

No major anticipated illness or organ failure incompatible with survival from BMT.

DLCO must not be less than 65% predicted.

No left ventricular ejection fraction: less than 40% predicted.

Must not have serum creatinine greater than 3 mg/dl.

Must not have serum bilirubin greater than 4 mg/dl, Transaminases greater than 3 times the upper limit of normal.

Donor or patient must not be HIV positive.

Must not have history of other malignancies except basal cell or squamous carcinoma of the skin, positive PAP smear and subsequent negative follow up.

Donor must be fit to receive G-CSF and undergo apheresis.

Must not fail to mobilize adequate numbers of CD34+ cells after two cycles of G-CSF.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35
Dates: Start 1998-06; Study Completion 2000-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Lane TA, Law P, Maruyama M, Young D, Burgess J, Mullen M, Mealiffe M, Terstappen LW, Hardwick A, Moubayed M, et al. Harvesting and enrichment of hematopoietic progenitor cells mobilized into the peripheral blood of normal donors by granulocyte-macrophage colony-stimulating factor (GM-CSF) or G-CSF: potential role in allogeneic marrow transplantation. Blood. 1995 Jan 1;85(1):275-82. PMID 7528570